CLINICAL TRIAL: NCT00323843
Title: RIRS - A Method of Treating the ESWL Resistant Kidney Stone
Brief Title: Retrograde Intrarenal Stone Surgery - A Method of Treating the ESWL Resistant Kidney Stone
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fredericia Hosptial (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-005972-34
Record Dates: First submitted 2006-05-08; First posted 2006-05-10 (Estimated); Last update posted 2007-01-30 (Estimated); Status verified 2007-01

CONDITIONS: Kidney Stone; Ureteroscopy
Keywords: Kidney stone; ureteropyeloscopy; renal pelvic pressure
MeSH Terms: conditions — Kidney Calculi | interventions — Isoproterenol

INTERVENTIONS:
Drug: Isoproterenol

SUMMARY:
Is it possible to decrease the intrarenal pressure in the kidney during endoscopic management of kidney stone by topical administration of drugs? In order to secure fewer complications in ureteroscopic operations the pharmacological agent isoproterenol is tested on pigs and human to determine its potential of lowering intrarenal pressure.

ELIGIBILITY:
Inclusion Criteria:

* Indication for RIRS procedure
* Age > 18 years
* Normotensive
* Capable of understanding information given

Exclusion Criteria:

* Previous myocardiac infarct
* Daily use of alpha- og beta- blocking medicine og calcium antagonists
* Use of NSAID the last 2 days
* Stone in the ureter
* Declared
* Known malignant disease in urinary tract
* Bladder disease
* Nephrostomies inserted
* JJ-catheters inserted
* Prisoners
* Pregnant
* Nursing mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2006-06; Study Completion 2007-02

PRIMARY OUTCOMES:
Renal pelvic pressure

SECONDARY OUTCOMES:
Blood pressure
Pulse

CONTACTS AND LOCATIONS:
Overall Officials: Helene U Jung, Principal Investigator — Fredericia Hospital, Dpt. of Urology
Locations (1):
- Dpt. of Urology, Fredericia, Vejle Council, Denmark